CLINICAL TRIAL: NCT06465797
Title: Collecting Imaging Data From Standard-of-care Bronchoscopies for AI-development: a Prospective, Non-interventional Study (Using CE-marked Bronchoscopes)
Brief Title: Observational Bronchoscopy Video Data Collection Study With Adult Patients
Status: Completed | Type: Observational
Sponsor: Ambu A/S (Industry)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ambu A/S
Record Dates: First submitted 2024-06-10; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Lung Diseases; Lung Neoplasms; Lung Cancer; Lung Transplantation; Lung Diseases, Obstructive
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms; Lung Diseases, Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — No intervention will take place in this study, only image material will be captured from the standard-of-care bronchoscopy

SUMMARY:
The primary aim is to develop a software algorithm that has the capacity to detect the normal 18 anatomical structures of the lung by using the position of the scope during the bronchoscopy procedure and using existing bronchoscopy technology.

DETAILED DESCRIPTION:
A data collection of bronchoscopy videos from 100-150 patients are enrolled for getting image material of different lung anatomies, captured with CE-marked and FDA-approved Ambu bronchoscopes (Ambu® aScope™ 5 Broncho HD). No intervention will take place, only standard of care. All types of indications are enrolled. All patients were given oral and written information prior to participating, and signed consent was provided. No patient identifiable information is stored.

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for bronchoscopy of central airways as per standard of care
* Patients of 18 years or above

Exclusion Criteria:

* Lack of patient cooperation for bronchoscopy (e.g. patients with mental disorders, dysgnosia, psychological disorder)
* Patients unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults indicated for a bronchoscopy above 18 year is part of the population.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Number of bronchial segments accessed during bronchoscopy | 1 year
  Accurate procedure recordings by the bronchoscope of all 18 anatomical segments +/- abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
The data is collected to develop software, and no intervention will take place. It will therefore not be relevant to share the data with other researchers for further analysis.